CLINICAL TRIAL: NCT00338117
Title: A European Multi-Center Study to Determine the Safety and Efficacy of Galanthamine Hydrobromide 40mg/Day (32 mg /Day GAL Base, Tid Dose Regimen) in Patients Diagnosed With Alzheimer-Type Dementia
Brief Title: Safety and Efficacy of High Dose, Rapid Titration Galantamine in Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Shire (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005884
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: Dementia; neurodegenerative disorder; impairment of memory; galantamine; galanthamine; acetylcholinesterase inhibitor; Mini Mental State Examination score
MeSH Terms: conditions — Alzheimer Disease; Dementia; Neurodegenerative Diseases | interventions — Galantamine

INTERVENTIONS:
Drug: Galantamine hydrobromide

SUMMARY:
The purpose of this study was to determine the safety and effectiveness of a relatively high dose of galantamine, 32 mg /day in a three-times daily dosage, compared with placebo in treating patients with Alzheimer's disease.

DETAILED DESCRIPTION:
Alzheimer's disease is a progressive degenerative brain disorder that affects memory, as well as the ability to concentrate, reason, and think in abstract form. This study was designed to examine the effectiveness and safety of galantamine (galant.) hydrobromide at a relatively high dose, compared with treatment with placebo, in men and women with Alzheimer's disease. Approximately 600 patients were screened. This was a double-blind study, i.e., neither patients nor investigators knew what treatment was given. Before the start of the double-blind phase, each patient was randomly assigned to receive either galantamine hydrobromide or placebo (i.e., no active drug). The dose was increased weekly, at a higher rate than currently recommended in the label, until the stable daily dose of 32 mg galantamine was reached. All patients took their treatment (galantamine or placebo) 3 times a day. All patients who completed the blinded phase of the study were permitted to enter an open-label phase, in which the treatment was made known to both investigators and patients. During this additional 24-week phase, all patients received treatment with galantamine hydrobromide. The effectiveness of study treatment (galantamine hydrobromide or placebo) was assessed using several measures and included the Mini Mental State Examination (MMSE) score. The MMSE consists of 12 questions and tasks designed to assess severity of Alzheimer's disease. Additional measures included the European Alzheimer Disease Assessment Scale cognitive score (EURO-ADAS-cog), a Clinician's Interview Based Impression of Change (CIBIC) plus, and the Nurses' Observation Scale for Geriatric Patients (NOSGER). Safety and tolerability were assessed using physical (full and brief) examination, adverse events reports, clinical and laboratory measures, and 12-lead ECG results. Galant. was taken orally as a tablet 3 times a day with meals. Patients started their treatment with a total 8 mg of galantamine. The dose was increased weekly to a daily cumulative dose of 32 mg (the same as 40 mg Gal HBr).This dose was higher and the titration schedule was 4 times more rapid that the 16 mg and 24 mg maintenance doses and 4-weekly titration steps specified in the US label. Each phase had a 5-week titration period. After 5 weeks, patients continued to receive 40 mg.

ELIGIBILITY:
Inclusion Criteria:

* Have been meeting the diagnostic criteria of Alzheimer's disease
* mild or moderate dementia as measured by the Mini Mental State Examination (MMSE) score
* live with or have daily visits from a responsible caregiver.

Exclusion Criteria:

* Parkinson's disease
* Pick's disease
* secondary or pseudodementias
* currently diagnosed epilepsy
* history of endocrine disorder
* significant heart disease
* drug or alcohol abuse
* kidney or liver dysfunction
* women of child-bearing potential unless appropriate birth-control method is used
* sensitivity to the study drug.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 1995-08; Study Completion 1997-05 (Actual)

PRIMARY OUTCOMES:
The primary outcomes included evaluations by EURO-ADAS cognitive score, CIBIC Plus, and NOSGER at 6 months.

SECONDARY OUTCOMES:
EURO-ADAS non-cognitive score; MMSE; Short Cognitive Performance Test (SKT) sub-set 6; Neuropsychological Assessment Battery (NAB); incidence of adverse events, changes in laboratory measures, results of physical exams, and results of 12-lead ECG.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.